CLINICAL TRIAL: NCT01336738
Title: A 12-Week, Phase 2, Randomized, Double-Blind, Placebo Controlled, Dose-Ranging, Parallel Group Study To Evaluate The Efficacy And Safety Of Once Daily Pf-04991532 And Sitagliptin In Adult Patients With Type 2 Diabetes Mellitus Inadequately Controlled On Metformin
Brief Title: Study Of Safety And Efficacy Of PF-04991532 In Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2611002
Record Dates: First submitted 2011-04-13; First posted 2011-04-18 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes, Type 2
Keywords: Phase 2; safety and efficacy study with PF-04991532; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Matching placebo for PF-04991532 and Sitagliptin
  Interventions: Drug: Placebo
- 150 mg PF-04991532 (Experimental)
  Interventions: Drug: 150 mg PF-04991532
- 450 mg PF-04991532 (Experimental)
  Interventions: Drug: 450 mg PF-04991532
- 750 mg PF-04991532 (Experimental)
  Interventions: Drug: 750 mg PF-04991532
- Sitagliptin 100 mg (Active Comparator)
  Interventions: Drug: Sitagliptin 100 mg

INTERVENTIONS:
Drug: Placebo — Tablets (n=6), 0 mg, once daily for 84 days
  Arms: Placebo
Drug: 150 mg PF-04991532 — Tablets (n=1), 150 mg + tablets (n=5), 0 mg, all once daily for 84 days
  Arms: 150 mg PF-04991532
Drug: 450 mg PF-04991532 — Tablets (n=3), 150 mg + tablets (n=3), 0 mg, all once daily for 84 days
  Arms: 450 mg PF-04991532
Drug: 750 mg PF-04991532 — Tablets (n=5), 150 mg + tablets (n=1), 0 mg, all once daily for 84 days
  Arms: 750 mg PF-04991532
Drug: Sitagliptin 100 mg — Tablets (n=1), 100 mg strength + tablets (n=5), 0 mg, all once daily for 84 days
  Arms: Sitagliptin 100 mg

SUMMARY:
B2611002 is designed to study how safe and effective an investigational medication (PF-04991532) is in people with Type 2 diabetes. Subjects in the study will receive 1 of 5 treatments for 3 months. One of the treatments will be sitagliptin which is an approved drug, and another treatment will be placebo, which does not contain active ingredient.

ELIGIBILITY:
Inclusion Criteria:

Subjects with type 2 diabetes on stable doses of background medicines for management of diabetes; aged 18-70 years; body mass index between 22.5 and 45.5 kg/m2

Exclusion Criteria:

Subjects with type 1 diabetes, heart attack or stroke in the past 6 months, uncontrolled blood pressure, significant kidney disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (24):
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Kenosha, Wisconsin
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Canada (6):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Strathroy, Ontario
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Saint Romuald, Quebec
- Pfizer Investigational Site, Budapest, Hungary
- Mexico (2):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Pfizer Investigational Site, Bratislava, Slovakia
- Pfizer Investigational Site, Seoul, South Korea
- Taiwan (2):
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611002&StudyName=Study%20Of%20Safety%20And%20Efficacy%20Of%20PF-04991532%20In%20Subjects%20With%20Type%202%20Diabetes%20Mellitus

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received placebo matched to PF-04991532 or placebo matched to sitagliptin tablet orally once daily along with background metformin immediate release tablets, during the 2-week run-in period. Compliant participants were then randomized to study treatments for 12 weeks.
Groups:
- PF-04991532 150 mg: PF-04991532 150 milligram (mg) (1 PF-04991532 150 mg tablet and 4 placebo tablets matched to PF-04991532 150 mg) orally once daily and 1 placebo tablet matched to sitagliptin 100 mg orally once daily, along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- PF-04991532 450 mg: PF-04991532 450 mg (3 PF-04991532 150 mg tablets and 2 placebo tablets matched to PF-04991532 150 mg) orally once daily and 1 placebo tablet matched to sitagliptin 100 mg orally once daily, along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- PF-04991532 750 mg: PF-04991532 750 mg (5 PF-04991532 150 mg tablets) orally once daily and 1 placebo tablet matched to sitagliptin 100 mg orally once daily, along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- Sitagliptin 100 mg: Five placebo tablets matched to PF-04991532 150 mg and 1 sitagliptin 100 mg tablet orally once daily, along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
- Placebo: Five placebo tablets matched to PF-04991532 150 mg and 1 placebo matched to sitagliptin 100 mg tablet orally once daily, along with background metformin 500 mg immediate release tablets or as per standard clinical practice (based on the dose prior to randomization), for 12 weeks.
Period: Overall Study
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Started | 52 | 54 | 53 | 54 | 53
Completed | 45 | 45 | 45 | 47 | 43
Not Completed | 7 | 9 | 8 | 7 | 10
Not completed — Adverse Event | 0 | 3 | 2 | 1 | 3
Not completed — Lost to Follow-up | 2 | 1 | 2 | 2 | 2
Not completed — Did not meet entrance criteria | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 1 | 1
Not completed — Other | 3 | 3 | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo | Total
Number analyzed (Participants) | 52 | 54 | 53 | 54 | 53 | 266
Age Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.9) | 55.1 (9.3) | 55.5 (7.3) | 57.8 (8.3) | 55.6 (8.5) | 55.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 24 | 17 | 23 | 14 | 94
  Male | 36 | 30 | 36 | 31 | 39 | 172

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. The normal range for the HbA1c test is between 4 percent (%) and 5.6%. HbA1c levels between 5.7% and 6.4% indicate increased risk of diabetes and levels of 6.5% or higher indicate diabetes.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication. Here 'n' signifies participants who were evaluable at specific time point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 52 | 53 | 52 | 54 | 53
percentage of hemoglobin
  Baseline (n=52, 53, 52, 54, 53) | 8.34 (0.906) | 8.19 (0.947) | 7.96 (1.030) | 7.97 (1.086) | 8.55 (1.351)
  Change at Week 12 (n=44, 44, 43, 48, 43) | -0.17 (0.922) | -0.57 (0.753) | -0.70 (0.790) | -0.78 (0.721) | -0.21 (0.921)
Statistical Analysis 1: Comparison: PF-04991532 150 mg vs Placebo; Treatment difference and 80% confidence interval (CI) were based on LS mean. A mixed model repeated measure (MMRM) analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.6803, Mixed Models Analysis — One-sided p-value was calculated; Least Squares (LS) Mean Difference = 0.08, 80% CI 2-sided [-0.13 to 0.29], Standard Error of Mean 0.164
Statistical Analysis 2: Comparison: PF-04991532 450 mg vs Placebo; Treatment difference and 80% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.49, 80% CI 2-sided [-0.71 to -0.28], Standard Error of Mean 0.166
Statistical Analysis 3: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.58, 80% CI 2-sided [-0.80 to -0.36], Standard Error of Mean 0.168
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.71, 80% CI 2-sided [-0.91 to -0.50], Standard Error of Mean 0.162

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 1, 2, 4, 8 and 12
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here 'n' signifies participants who were evaluable at specific time point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 52 | 53 | 52 | 54 | 53
milligram/deciliter (mg/dL)
  Baseline (n=52, 53, 52, 54, 53) | 172.68 (39.612) | 169.16 (41.703) | 159.11 (44.878) | 158.38 (42.502) | 183.61 (57.517)
  Change at Week 1 (n=50, 51, 49, 49, 51) | 0.87 (27.059) | 1.63 (25.373) | -1.55 (19.826) | -13.72 (24.445) | -4.21 (33.274)
  Change at Week 2 (n=50, 51, 51, 50, 47) | -4.48 (23.488) | 4.13 (30.662) | -5.26 (21.466) | -15.70 (29.704) | -3.72 (27.797)
  Change at Week 4 (n=49, 49, 49, 50, 45) | 1.13 (28.589) | -5.14 (29.757) | -6.68 (20.582) | -21.86 (29.063) | -4.28 (34.304)
  Change at Week 8 (n=46, 44, 44, 47, 45) | 3.69 (29.232) | -1.49 (33.421) | 2.95 (21.892) | -14.05 (21.646) | 2.18 (37.322)
  Change at Week 12 (n=45, 44, 44, 48, 43) | 0.08 (36.122) | 5.87 (33.092) | 6.86 (28.602) | -17.64 (30.779) | -0.03 (45.784)
Statistical Analysis 1: Comparison: PF-04991532 150 mg vs Placebo; Week 1: Treatment difference and 95% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.4757, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 3.78, 95% CI 2-sided [-6.64 to 14.20], Standard Error of Mean 5.292
Statistical Analysis 2: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8031, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 1.32, 95% CI 2-sided [-9.11 to 11.75], Standard Error of Mean 5.296
Statistical Analysis 3: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5490, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -3.22, 95% CI 2-sided [-13.78 to 7.34], Standard Error of Mean 5.364
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -15.07, 95% CI 2-sided [-25.58 to -4.55], Standard Error of Mean 5.340
Statistical Analysis 5: Comparison: PF-04991532 150 mg vs Placebo; Week 2: Treatment difference and 95% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.6291, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -2.43, 95% CI 2-sided [-12.31 to 7.46], Standard Error of Mean 5.020
Statistical Analysis 6: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.4396, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 3.87, 95% CI 2-sided [-5.98 to 13.72], Standard Error of Mean 5.001
Statistical Analysis 7: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.1934, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -6.56, 95% CI 2-sided [-16.46 to 3.34], Standard Error of Mean 5.030
Statistical Analysis 8: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -17.32, 95% CI 2-sided [-27.24 to -7.40], Standard Error of Mean 5.039
Statistical Analysis 9: Comparison: PF-04991532 150 mg vs Placebo; Week 4: Treatment difference and 95% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.5479, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 3.13, 95% CI 2-sided [-7.11 to 13.37], Standard Error of Mean 5.201
Statistical Analysis 10: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.4276, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -4.14, 95% CI 2-sided [-14.39 to 6.12], Standard Error of Mean 5.209
Statistical Analysis 11: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.1596, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -7.38, 95% CI 2-sided [-17.69 to 2.92], Standard Error of Mean 5.235
Statistical Analysis 12: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -22.83, 95% CI 2-sided [-33.06 to -12.60], Standard Error of Mean 5.198
Statistical Analysis 13: Comparison: PF-04991532 150 mg vs Placebo; Week 8: Treatment difference and 95% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.8509, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -1.10, 95% CI 2-sided [-12.63 to 10.43], Standard Error of Mean 5.855
Statistical Analysis 14: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.1505, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -8.53, 95% CI 2-sided [-20.17 to 3.12], Standard Error of Mean 5.913
Statistical Analysis 15: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.2662, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -6.62, 95% CI 2-sided [-18.31 to 5.08], Standard Error of Mean 5.940
Statistical Analysis 16: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -21.52, 95% CI 2-sided [-32.97 to -10.07], Standard Error of Mean 5.818
Statistical Analysis 17: Comparison: PF-04991532 150 mg vs Placebo; Week 12: Treatment difference and 95% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.7724, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -2.01, 95% CI 2-sided [-15.68 to 11.66], Standard Error of Mean 6.940
Statistical Analysis 18: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.9202, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -0.70, 95% CI 2-sided [-14.47 to 13.07], Standard Error of Mean 6.986
Statistical Analysis 19: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.8183, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -1.61, 95% CI 2-sided [-15.40 to 12.18], Standard Error of Mean 6.998
Statistical Analysis 20: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -24.96, 95% CI 2-sided [-38.40 to -11.53], Standard Error of Mean 6.821

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 1, 2, 4 and 8
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. The normal range for the HbA1c test is between 4% and 5.6%. HbA1c levels between 5.7% and 6.4% indicate increased risk of diabetes and levels of 6.5% or higher indicate diabetes.
Time Frame: Baseline, Week 1, 2, 4, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 52 | 53 | 52 | 54 | 53
percentage of hemoglobin
  Change at Week 1 (n=50, 51, 49, 49, 48) | -0.04 (0.227) | -0.03 (0.210) | -0.13 (0.217) | -0.07 (0.200) | -0.02 (0.287)
  Change at Week 2 (n=50, 52, 49, 49, 47) | -0.04 (0.349) | -0.14 (0.288) | -0.18 (0.271) | -0.23 (0.311) | -0.07 (0.372)
  Change at Week 4 (n=48, 49, 48, 50, 46) | -0.22 (0.475) | -0.34 (0.392) | -0.40 (0.421) | -0.42 (0.483) | -0.16 (0.591)
  Change at Week 8 (n=45, 44, 45, 47, 45) | -0.21 (0.728) | -0.50 (0.562) | -0.66 (0.772) | -0.71 (0.713) | -0.22 (0.762)
Statistical Analysis 1: Comparison: PF-04991532 150 mg vs Placebo; Week 1: Treatment difference and 80% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.2327, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.04, 80% CI 2-sided [-0.10 to 0.03], Standard Error of Mean 0.048
Statistical Analysis 2: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3580, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.02, 80% CI 2-sided [-0.08 to 0.04], Standard Error of Mean 0.048
Statistical Analysis 3: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0036, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.13, 80% CI 2-sided [-0.20 to -0.07], Standard Error of Mean 0.049
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1251, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.06, 80% CI 2-sided [-0.12 to 0.01], Standard Error of Mean 0.049
Statistical Analysis 5: Comparison: PF-04991532 150 mg vs Placebo; Week 2: Treatment difference and 80% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.3466, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.03, 80% CI 2-sided [-0.11 to 0.06], Standard Error of Mean 0.066
Statistical Analysis 6: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.0439, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.11, 80% CI 2-sided [-0.20 to -0.03], Standard Error of Mean 0.066
Statistical Analysis 7: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.0040, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.18, 80% CI 2-sided [-0.27 to -0.09], Standard Error of Mean 0.067
Statistical Analysis 8: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.20, 80% CI 2-sided [-0.29 to -0.12], Standard Error of Mean 0.065
Statistical Analysis 9: Comparison: PF-04991532 150 mg vs Placebo; Week 4: Treatment difference and 80% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.1405, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.10, 80% CI 2-sided [-0.23 to 0.02], Standard Error of Mean 0.096
Statistical Analysis 10: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.0067, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.24, 80% CI 2-sided [-0.36 to -0.12], Standard Error of Mean 0.097
Statistical Analysis 11: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.37, 80% CI 2-sided [-0.50 to -0.24], Standard Error of Mean 0.098
Statistical Analysis 12: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.34, 80% CI 2-sided [-0.46 to -0.22], Standard Error of Mean 0.094
Statistical Analysis 13: Comparison: PF-04991532 150 mg vs Placebo; Week 8: Treatment difference and 80% CI were based on LS mean. A MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, baseline-by-time interaction as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.4887, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = 0.00, 80% CI 2-sided [-0.18 to 0.17], Standard Error of Mean 0.135
Statistical Analysis 14: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.40, 80% CI 2-sided [-0.57 to -0.22], Standard Error of Mean 0.137
Statistical Analysis 15: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.58, 80% CI 2-sided [-0.76 to -0.41], Standard Error of Mean 0.138
Statistical Analysis 16: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — One-sided p-value was calculated; LS Mean Difference = -0.59, 80% CI 2-sided [-0.76 to -0.42], Standard Error of Mean 0.133

4. Secondary Outcome: Percentage of Participants Achieving Less Than (<) 6.5% or <7% Glycosylated Hemoglobin (HbA1c) Levels
Description: as for outcome 3
Time Frame: Week 12
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, N (number of participants analyzed) signify those who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 44 | 44 | 43 | 48 | 43
percentage of participants
  < 6.5% | 4.5 | 9.1 | 23.3 | 14.6 | 11.6
  < 7% | 13.6 | 36.4 | 60.5 | 39.6 | 16.3

5. Secondary Outcome: Change From Baseline in Body Weight at Week 1, 2, 4, 8 and 12
Description: Overweight or obesity increases the risk for developing diabetes. The treatment of diabetes has been the recommendation to lose weight. As weight loss progresses and is maintained, an improvement of glycemia may be evidenced by a reduction in HbA1c.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 52 | 53 | 52 | 54 | 53
kilogram (kg)
  Baseline (n=52, 53, 52, 54, 53) | 92.57 (19.957) | 88.91 (22.781) | 86.08 (17.787) | 87.48 (19.883) | 87.43 (19.351)
  Change at Week 1 (n=50, 51, 49, 51, 51) | -0.10 (1.176) | -0.31 (1.091) | -0.34 (1.100) | 0.14 (0.982) | -0.33 (1.050)
  Change at Week 2 (n=50, 52, 51, 50, 48) | -0.12 (1.189) | -0.33 (1.175) | -0.38 (1.115) | -0.00 (1.364) | -0.37 (0.885)
  Change at Week 4 (n=49, 49, 49, 50, 46) | -0.18 (1.357) | -0.72 (1.499) | -0.34 (1.486) | 0.15 (1.170) | -0.52 (1.139)
  Change at Week 8 (n=46, 44, 45, 48, 45) | -0.27 (1.865) | -0.66 (2.047) | -0.45 (2.026) | -0.21 (2.059) | -0.60 (1.444)
  Change at Week 12 (n=45, 44, 45, 48, 43) | -0.91 (1.880) | -0.82 (2.126) | -0.90 (2.421) | -0.22 (1.993) | -0.95 (2.058)
Statistical Analysis 1: Comparison: PF-04991532 150 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2067, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.28, 95% CI 2-sided [-0.16 to 0.73], Standard Error of Mean 0.225
Statistical Analysis 2: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8602, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.04, 95% CI 2-sided [-0.40 to 0.48], Standard Error of Mean 0.224
Statistical Analysis 3: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9200, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -0.02, 95% CI 2-sided [-0.47 to 0.42], Standard Error of Mean 0.225
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0399, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.46, 95% CI 2-sided [0.02 to 0.90], Standard Error of Mean 0.223
Statistical Analysis 5: Comparison: PF-04991532 150 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.2266, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.29, 95% CI 2-sided [-0.18 to 0.77], Standard Error of Mean 0.242
Statistical Analysis 6: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.8493, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.05, 95% CI 2-sided [-0.43 to 0.52], Standard Error of Mean 0.241
Statistical Analysis 7: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.9511, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -0.01, 95% CI 2-sided [-0.49 to 0.46], Standard Error of Mean 0.242
Statistical Analysis 8: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.1369, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.36, 95% CI 2-sided [-0.11 to 0.83], Standard Error of Mean 0.241
Statistical Analysis 9: Comparison: PF-04991532 150 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.1562, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.39, 95% CI 2-sided [-0.15 to 0.92], Standard Error of Mean 0.272
Statistical Analysis 10: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.4913, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -0.19, 95% CI 2-sided [-0.72 to 0.35], Standard Error of Mean 0.272
Statistical Analysis 11: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.5130, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.18, 95% CI 2-sided [-0.36 to 0.71], Standard Error of Mean 0.272
Statistical Analysis 12: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.0298, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.59, 95% CI 2-sided [0.06 to 1.12], Standard Error of Mean 0.269
Statistical Analysis 13: Comparison: PF-04991532 150 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.3196, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.36, 95% CI 2-sided [-0.35 to 1.08], Standard Error of Mean 0.363
Statistical Analysis 14: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.8884, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = -0.05, 95% CI 2-sided [-0.77 to 0.67], Standard Error of Mean 0.367
Statistical Analysis 15: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.7325, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.12, 95% CI 2-sided [-0.59 to 0.84], Standard Error of Mean 0.365
Statistical Analysis 16: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 13]; Test type: Superiority or Other; p = 0.3395, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.34, 95% CI 2-sided [-0.36 to 1.04], Standard Error of Mean 0.357
Statistical Analysis 17: Comparison: PF-04991532 150 mg vs Placebo; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.7514, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.13, 95% CI 2-sided [-0.68 to 0.94], Standard Error of Mean 0.410
Statistical Analysis 18: Comparison: PF-04991532 450 mg vs Placebo; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.7529, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.13, 95% CI 2-sided [-0.68 to 0.94], Standard Error of Mean 0.413
Statistical Analysis 19: Comparison: PF-04991532 750 mg vs Placebo; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.9638, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.02, 95% CI 2-sided [-0.79 to 0.83], Standard Error of Mean 0.411
Statistical Analysis 20: Comparison: Sitagliptin 100 mg vs Placebo; [analysis description as in outcome 2, analysis 17]; Test type: Superiority or Other; p = 0.0962, Mixed Models Analysis — Two-sided p-value was calculated; LS Mean Difference = 0.67, 95% CI 2-sided [-0.12 to 1.47], Standard Error of Mean 0.404

6. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 1% or >= 2% Body Weight Gain From Baseline
Description: Overweight or obesity increases the risk for developing diabetes. Participants with >= 1% or >= 2% body weight gain from baseline signifies a higher risk of diabetes.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 45 | 44 | 45 | 48 | 43
percentage of participants
  >= 1% | 17.78 | 18.18 | 15.56 | 29.17 | 23.26
  >= 2% | 6.67 | 11.36 | 11.11 | 14.58 | 6.98

7. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 1% or >= 2% Body Weight Loss From Baseline
Description: The treatment of diabetes has been the recommendation to lose weight. As weight loss progresses and is maintained, an improvement of glycemia may be evidenced by a reduction in HbA1c. Participants with >= 1% or >= 2% body weight loss from baseline signifies an improvement of glycemia.
Time Frame: Week 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 45 | 44 | 45 | 48 | 43
percentage of participants
  >= 1% | 55.56 | 47.73 | 46.67 | 29.17 | 41.86
  >= 2% | 26.67 | 34.09 | 31.11 | 18.75 | 34.88

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04991532 150 mg | PF-04991532 450 mg | PF-04991532 750 mg | Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/54 | 0/53 | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 17/52 | 20/54 | 23/53 | 14/54 | 16/53
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04991532 150 mg (N=52) | PF-04991532 450 mg (N=54) | PF-04991532 750 mg (N=53) | Sitagliptin 100 mg (N=54) | Placebo (N=53)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 7 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 4 | 2 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1
Influenza (Infections and infestations) | 2 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 3 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 3 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2
Hypertension (Vascular disorders) | 0 | 3 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.